CLINICAL TRIAL: NCT06646081
Title: The Effects of Greater Occipital Nerve and Stellate Ganglion Blocks on Sleep Quality in Chronic Headache Patients: A Randomized Controlled Trial
Brief Title: The Impact of Greater Occipital Nerve and Stellate Ganglion Block Treatments on Sleep in Chronic Headache Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Turan, MD, Principal Investigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GON block vs Stellate block
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Chronic Headache; Chronic Headache Disorder; Migraine
Keywords: stellate ganglion block; greater occipital nerve block
MeSH Terms: conditions — Headache Disorders; Migraine Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greater Occipital Nerve Block Group (Active Comparator): Greater Occipital Nerve Block for Chronic Headache
  Interventions: Procedure: Greater Occipital Nerve Block
- Stellate Ganglion Block Group (Active Comparator): Stellate Ganglion Block for Chronic Headache
  Interventions: Procedure: Stellate Ganglion Block

INTERVENTIONS:
Procedure: Greater Occipital Nerve Block — The patient is placed prone with the head neutral or slightly flexed. After sterile preparation, a high-frequency linear probe is positioned transversely at the upper nuchal line in the occipital region. The Greater Occipital Nerve, exiting from the posterior root of C2, is located near the occipital artery. Using an in-plane technique, a 25-gauge needle is inserted into the fascial plane around the artery. After confirming no intravascular placement by negative aspiration, 5 mL of a mixture of 50 mg lidocaine and isotonic saline is injected. The fascial plane opening confirms the site. The area is dressed, and the patient is monitored for one hour for side effects.
  Arms: Greater Occipital Nerve Block Group
Procedure: Stellate Ganglion Block — The patient lies supine with a pillow under the shoulders, and the head slightly extended, neck gently turned opposite to the blockade. After sterile preparation, a high-frequency linear probe is placed transversely at the C6 vertebra (Chassaignac's tubercle). Ultrasound identifies the C6 vertebra, Longus colli muscle, carotid artery, and internal jugular vein. The Stellate Ganglion is located within the prevertebral fascia over the Longus colli. Using an in-plane technique, a 25-gauge needle is inserted and advanced into the prevertebral fascial plane. After confirming no intravascular placement by negative aspiration, 5 mL of 50 mg lidocaine and isotonic saline is injected. The fascial plane opening confirms the site. The area is dressed, and the patient is monitored for one hour for side effects.
  Arms: Stellate Ganglion Block Group

SUMMARY:
This study aims to evaluate the effect of Greater Occipital Nerve and Stellate Ganglion block treatments on sleep in patients with chronic headaches. Patients will be assessed using the Pittsburgh Sleep Quality Index, Insomnia Severity Index, and Visual Analog Scale at the time of treatment and at 4 and 8 weeks post-procedure. The study will compare the sleep improvement effects of both treatments to help guide clinicians in selecting the most effective interventional method. Demographic and clinical data will also be collected and analyzed for statistical comparison.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of Greater Occipital Nerve and Stellate Ganglion blockade treatments, used in the treatment of chronic headache, on sleep. These treatments were administered in two sessions, one week apart, for chronic headache. The goal is to compare the treatments using scales at the time of application and at the fourth and eighth weeks after the last procedure.

The improvement effect of Greater Occipital Nerve block on sleep quality scales has recently been reported in several studies in the literature. However, the efficacy of Stellate Ganglion block, a proven method for headache treatment, in these areas has not yet been studied, and its effect on sleep improvement will be investigated.

It is believed that determining the superiority of the interventional methods used on sleep, based on scales, will assist clinicians in decision-making when performing the procedure.

Patients with chronic headache (lasting more than 3 months) who undergo Greater Occipital Nerve or Stellate Ganglion blockade at the clinic will be evaluated. The Pittsburgh Sleep Quality Index and Insomnia Severity Index will be applied immediately after the procedure and at the 4th and 8th weeks following the last procedure. The Visual Analog Scale (VAS) will be obtained from clinic notes for the pre-procedure value and will be repeated at the 4th and 8th weeks post-procedure. The administration of scales will be conducted at Etlik City Hospital Algology Clinic. Patients will be evaluated either during outpatient follow-up or by phone. This study will not include sensitive or vulnerable patient groups. Demographic characteristics (age, gender, height, weight, BMI, alcohol, and smoking habits), comorbidities (obesity, restless legs, psychiatric disorders, sleep disorders, medications), and the scores from the mentioned scales will be recorded and statistically compared.

ELIGIBILITY:
Inclusion Criteria:

* Chronic headache unresponsive to conservative treatment
* Male and female population aged 18-50
* No prior interventional procedures during the treatment process

Exclusion Criteria:

* Coagulation disorders
* Infections at the procedure site
* Allergy to local anesthesia
* Socio-cultural inadequacy
* Mental retardation
* Pregnancy
* Previous interventional procedures
* Patient refusal of interventional procedure
* Use of any sleep-improving medication within the last month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Change from baseline to 1st and 2nd month after treatment
  The Pittsburgh Sleep Quality Index is a questionnaire designed to assess sleep quality and disturbances over a one-month period. It consists of 19 self-rated questions and 5 questions rated by a bed partner or roommate (if available), which are not included in the score. The Pittsburgh Sleep Quality Index generates seven component scores, which are combined to produce a global score ranging from 0 to 21, with higher scores indicating worse sleep quality. A score greater than 5 indicates poor sleep quality.assess sleep quality and disturbances over a one-month period.
Insomnia Severity Index | Change from baseline to 1st and 2nd month after treatment
  The Insomnia Severity Index is a self-reported questionnaire designed to assess the severity of insomnia symptoms and their impact on daily functioning. The Insomnia Severity Index consists of 7 items that assess the severity of sleep onset, sleep maintenance difficulties, early morning awakenings, satisfaction with sleep, interference with daily functioning, noticeability of impairment attributed to sleep problems, and the level of distress caused by sleep difficulties. The total Insomnia Severity Index score ranges from 0 to 28, with higher scores indicating more severe insomnia.

SECONDARY OUTCOMES:
Numeric Rating Scale | Change from baseline to 1st and 2nd month after treatment
  Numeric Rating Scale is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioglu, Study Chair — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Etlik, Turkey (Türkiye)